CLINICAL TRIAL: NCT01752244
Title: Assessing the Effects of Supplementary Alfacalcidol Intake on Peroxisome Proliferator-activated Receptor-coactivator-1α, Vitamin D Receptor and Peroxisome Proliferator-activated Receptor Gamma Gene Expression in Obese Subjects
Brief Title: Assessing the Effects of Alfacalcidol Intake on Expression of Involed Gene in Metabolism in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91-02-27-18041
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Obesity
Keywords: Obesity, vitamin D analogue, VDR, PPARg, PGC1a
MeSH Terms: conditions — Obesity; Carotid Intimal Medial Thickness 1 | interventions — Corn Oil; alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Alfacalcidol (Experimental): Alfacalcidol
  Interventions: Dietary Supplement: Alfacalcidol
- Placebo (Placebo Comparator): Corn oil pearl Capsules 1 gram: were given to the intervention group once a day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — corn oil Capsules 1 gram: were given to the placebo group once a day for 8 weeks
  Other Names: corn oil capsule; Corn oil Pearl
  Arms: Placebo
Dietary Supplement: Alfacalcidol — Alfacalcidol
  Other Names: One-Alpha® Capsules 1 microgram; 1-α hydroxyvitamin D3
  Arms: Alfacalcidol

SUMMARY:
Obesity-induced chronic inflammation is a key component of the pathogenesis of insulin resistance. Mounting evidence has demonstrated anti-inflammatory characteristics for vitamin D. Although analogues of vitamin D3 have extensively been used in the treatment of various chronic inflammatory diseases, to our knowledge, no such research is conducted in regards with obesity. The aim of this double blind clinical trial study is to investigate whether alphacalcidol treatment in obese subjects can affect the insulin resistance. Moreover, we will evaluate the pathways of Vitamin D receptor (VDR), Peroxisome proliferator-activated receptor gamma (PPARγ) and eroxisome proliferator-activated receptor- coactivator-1 α (PGC1α) gene expressions which may lead to insulin resistance following treatment with either alphacalcidol or placebo.

DETAILED DESCRIPTION:
Increasing evidence from human population studies and animal research has established correlative as well as causative links between chronic inflammation and insulin resistance. The anti-inflammatory characteristics of vitamin D have been demonstrated in previous studies. In addition to its role in bone and calcium metabolism, vitamin D is demonstrated to be influential in the regulation of different immune system functions and glucose homeostasis pathways. Although low levels of vitamin D have shown to be in close correlation with obesity, whether vitamin D deficiency is the cause or the consequence of obesity remains unclear. It is noteworthy that several studies have demonstrated that vitamin D deficiency is associated with an increased resistance to insulin.

The biologic effects of vitamin D are primarily mediated via the nuclear transcription factor, vitamin D receptor (VDR), which triggers the expression of vitamin D responsive genes. VDR is expressed on different immune cells such as monocytes, T-lymphocytes, and granulocytes. It is documented that VDR and PGC-1α show an overlapping pattern of expression. Furthermore, as the expression of PGC-1α and PPARγ are regulated via environmental stimuli such as diet, it could be suggested that the function of VDR function can also be altered in response to external stimuli. PGC-1α was demonstrated to be of a particular importance in amelioration of increased insulin sensitivity.

Accordingly, to evaluate whether alphacalcidol treatment in obese subjects who generally suffer from a low state chronic inflammation could affect the insulin resistance, we designed the current double blind clinical trial study to compare the effect of alfacalcidol with placebo on serum glucose, 25-OH vitamin D, PTH, and lipid profile levels as well as Homeostatic model assessment (HOMA) and quantitative insulin sensitivity check index (QUICKI) indexes as a markers of insulin resistance. Furthermore, to assess the possible cross talk between VDR and PPARγ, the gene expressions of these VDR, PPARγ and PGC1α were evaluated following a course of treatment with either alphacalcidol or placebo.

ELIGIBILITY:
Inclusion Criteria:

Age 22-52 years Body mass index equal or more than 30

Exclusion criteria:

Acute or chronic inflammatory disease History of hypertension Alcohol or drug abuse History of any condition affecting inflammatory markers such as known cardiovascular disease Thyroid diseases Malignancies Current smoking Diabetes mellitus Sustained hypertension Heart failure Acute or chronic infections Hepatic or renal diseases Use of PPARγ agonist drug

Ages: 22 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Expression of VDR, PPARγ and PGC1α gene | Change from baseline to 8 weeks
  measurement of Relative gene expression with RT-PCR.

SECONDARY OUTCOMES:
Change of weight | Change from baseline to 8 weeks
  measurement with Body composition device

OTHER OUTCOMES:
Body mass index change | Change from baseline to 8 weeks
  calculated with BMI equation

CONTACTS AND LOCATIONS:
Overall Officials: Arash Hossein-nezhad, MD, PhD, Principal Investigator — Tehran University of Medical Sciences; Khadijeh Mirzaei, Ms, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- TehranUMS, Tehran, Iran

REFERENCES:
- [Derived] Mirzaei K, Hossein-Nezhad A, Keshavarz SA, Eshaghi SM, Koohdani F, Saboor-Yaraghi AA, Hosseini S, Tootee A, Djalali M. Insulin resistance via modification of PGC1alpha function identifying a possible preventive role of vitamin D analogues in chronic inflammatory state of obesity. A double blind clinical trial study. Minerva Med. 2014 Feb;105(1):63-78. PMID 24572452